CLINICAL TRIAL: NCT05493462
Title: A Clinical Research Study Evaluating the Safety, Tolerability and Efficacy of Intranasally Administered Human FGF-1 in Subjects With Parkinson's Disease
Brief Title: Intranasal Human FGF-1 for Subjects With Parkinson's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhittya Genesis Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MROS/457920/INDTP
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Human FGF-1 — Intranasal administration of human FGF-1

SUMMARY:
This is an open-label, pilot study to evaluate the safety, tolerability and efficacy of two dose levels of human FGF-1 administered intranasally to subjects with Parkinson's disease. A low dose of 450 µg FGF-1 (6 µg/kg for a 75 kg subject) and a high dose of 900 µg FGF-1 (12 µg/kg for a 75 kg subject) will be studied sequentially.

DETAILED DESCRIPTION:
The primary objectives of this study are to determine the safety, tolerability and efficacy of human fibroblast growth factor 1 (FGF-1) when administered intranasally to four (4) subjects with idiopathic, stage III or IV Parkinson's disease (Hoehn and Yahr staging criteria). This is an open-label, pilot study to study two dose levels of human FGF-1. A low dose of 450 µg FGF-1 (6 µg/kg for a 75 kg subject) and a high dose of 900 µg FGF-1 (12 µg/kg for a 75 kg subject) will be studied sequentially. Subjects will be screened up to 14 days before administration of the investigational drug product (FGF-1). If the subject complies with all inclusion/exclusion criteria, they will be enrolled in the study.

The proposed daily intranasal dosing regimen for the four subjects is as follows:

Week 1: 450 µg FGF-1 Week 2: 450 µg FGF-1 Week 3: No patient dosing, but safety and efficacy testing will be performed. If deemed safe, but a documented improvement in efficacy is not observed, the four subjects will proceed to administration of a higher dose of FGF-1.

Week 4: daily dosing with 900 µg FGF-1 Weeks 5-12: Follow-up weekly visits; no drug dosing; only safety and efficacy testing will be performed.

Prior to delivering the drug, the subject's vital signs will be taken. Following the intranasal delivery of the FGF-1 dose by the ViaNase® Electronic Atomizer (this device, which the U.S. FDA has authorized for use in humans, releases a metered dose of a drug into each nostril of the subject's nose, which then is inhaled by breathing evenly over a 2-minute period). Vital signs will be measured after the two-minute breathing period and then again in 15 minutes and 30 minutes. Following the final dosing period, follow-up visits for safety testing and efficacy evaluations will be given at weekly intervals for the following 7 weeks.

Safety and tolerability will be assessed by evaluating adverse events (AEs) (including a battery of laboratory evaluations, vital signs, physical examination findings, eye exams, and electrocardiograms [ECGs]). Efficacy will be assessed with the U.S. Movement Disorder Society-Sponsored Revision of the Uniﬁed Parkinson's Disease Rating Scale (MDS-UPDRS). This is a validated questionnaire that takes 30 minutes for a trained medical professional to administer to patients and measures the longitudinal progression of Parkinson's disease, including a section on motor skill testing.

Expected outcomes from this study include establishing that human FGF-1 is safe and tolerable when administered intranasally to subjects with Parkinson's disease and that a clinical benefit is observed in these patients, who currently have very limited medical options.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 40-80 years of age, inclusive, with a diagnosis of Parkinson's disease. At screening, a further confirmation of the diagnosis of Parkinson's disease will be made by the PI in accordance with accepted medical practices.
2. Female subjects of non-childbearing potential or if of child-bearing potential, on birth control deemed acceptable to the Principal Investigator (PI).
3. Signed and dated informed consent form, which meets all current regulatory criteria.
4. No evidence of proliferative retinopathy or significant non-proliferative retinopathy.
5. Subjects can be on a stable medical therapy for their Parkinson's disease prior to entering the study, as documented by their medical history. Other medications that are acceptable will be at the discretion of the Principal Investigator. At screening it will be stressed that, if possible, subjects should not add, switch or increase doses of any Parkinson's disease medications during the duration of the study.
6. Test drug administration and administration of questionnaires to measure motor function and mental status will be performed in the "on" state.
7. Ability to complete the study in compliance with the protocol in the opinion of the Principal Investigator.

   -

Exclusion Criteria:

1. Females who are pregnant at screening or of child-bearing potential and not using an acceptable form of birth control.
2. History of allergy or sensitivity to heparin.
3. Significant history or current evidence of chronic infectious disease or other medical conditions that, in the opinion of the Investigator, would compromise the safety of the subject or the study.
4. Subjects with malignancies or a history of malignancies (with the exception of basal cell carcinoma or squamous cell carcinoma of the skin) will be excluded from the study.
5. Clinically significant ECG abnormalities that in the opinion of the PI could potentially put the patient at risk.
6. Subjects with an HbA1C of >7.5%
7. Uncontrolled hypertension with systolic blood pressure >165 mmHg or diastolic blood pressure >100 mmHg despite diet, exercise or a stable dose of an appropriate antihypertensive therapy for at least 3 months
8. Significant hypotension with systolic blood pressure <85 mmHg or diastolic blood pressure <55 mmHg.
9. Total fasting serum cholesterol >220 mg/dL.
10. A current diagnosis or recent history of psychotic disorder, MDD, bipolar disorder, or posttraumatic stress disorder, or other psychiatric condition that, in the Investigator's opinion, would interfere with the subject's ability to participate in the trial.
11. Current use of tobacco products (may have a past history of tobacco use, but not in the last 3 months)
12. Pre-existing retinal disease, including proliferative retinopathy or severe nonproliferative retinopathy
13. Evidence suggesting any type of non-Parkinson disease movement disorder including progressive supranuclear palsy, multiple system atrophy, spinal cerebellar ataxia, etc.
14. Patients who are immunosuppressed.
15. Receipt of any drug as part of a research study within 3 months of the screening visit.
16. History of substance use disorder of moderate to severe severity within 3 months before screening or positive drugs of abuse testing on screening.
17. History of alcohol use disorder of moderate to severe severity within 6 months before screening requiring hospitalization or treatment at an inpatient treatment center.
18. Positive test results for HIV or hepatitis B and C antibodies.
19. Any abnormal laboratory value, condition, medication or medical device that in the opinion of the Principal Investigator could potentially compromise the patient's safety.
20. Unable or unwilling to make the required study visits -

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 12 weeks
  Adverse events

SECONDARY OUTCOMES:
Efficacy | 12 weeks
  Motor skill improvement by Parkinson's disease questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical Pavilion Bahamas, Nassau, The Bahamas

IPD SHARING:
Plan to Share IPD: No